CLINICAL TRIAL: NCT00585624
Title: Preoperative Nutritional Support Reduces Postoperative Stay and Incidence of Complications in Patients Undergoing an Esophagectomy or Pancreaticoduodenectomy
Brief Title: Preoperative Nutritional Support in Esophagectomy or Pancreaticoduodenectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 06206; #H-2006-0401
Record Dates: First submitted 2007-12-26; First posted 2008-01-03 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Esophagectomy; Pancreaticoduodenectomy
Keywords: Esophagectomy; Pancreaticoduodenectomy; Whipple

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Supplement: 3 servings/day of Impact Advanced Recovery in addition to regular food or any other supplements recommended or desired by patient or primary care/surgical team.
  Interventions: Dietary Supplement: Impact Advanced Recovery
- 2 (Placebo Comparator): Standard Care: Food, beverages, or supplements as recommended or desired by patient or primary care/surgical team.
  Interventions: Dietary Supplement: No supplement

INTERVENTIONS:
Dietary Supplement: Impact Advanced Recovery — Nutritional supplement
  Arms: 1
Dietary Supplement: No supplement — No supplement
  Arms: 2

SUMMARY:
We are proposing to evaluate the benefit of preoperative nutritional support with Impact Advanced Recovery in the most vulnerable group of elective gastrointestinal surgery patients who may experience a complication, esophagus and pancreas resections, and hypothesize that oral supplementation with 3 servings (0.75 L) Impact Advanced Recovery will reduce postoperative stay by 10-20% and reduce the incidence of major complications by 25%.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age 18 years or older of any race-ethnicity who will undergo an elective esophagectomy or pancreaticoduodenectomy.
2. Surgery will be scheduled 5-7 days after consent date -

Exclusion Criteria:

1. Surgery is urgent or emergent and/or patient would be unable to consume nutritional supplement for 5-7 days
2. Patient is currently receiving enteral (tube) or parenteral (IV) nutritional support
3. Patients with known pre-existing renal failure requiring a low protein diet
4. Patient is unable to drink 3 servings/day of a liquid supplement -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Estimated)
Dates: Start 2007-04; Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Postoperative stay in days | Postoperative stay in hospital & 30 days

SECONDARY OUTCOMES:
Incidence of major complications | Postoperative stay in hospital & 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth A Kudsk, MD, Principal Investigator — University of Wisconsin School of Medicine & Public Health
Locations (1):
- University of Wisconsin Hospital & Clinics, Madison, Wisconsin, United States